CLINICAL TRIAL: NCT06761469
Title: Pragmatic, Randomized, Cluster Stepped-Wedge Clinical Trial for Active Case Finding of Leprosy in Brazil
Brief Title: Leprosy Active Searching Trial in Brazil
Acronym: LAST•Br
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Alemão Oswaldo Cruz (Other)
Responsible Party: Principal Investigator, Sebastian Andres Vernal Carranza, Medical Doctor, Hospital Alemão Oswaldo Cruz
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 78510724.3.0000.0070
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Leprosy
Keywords: Leprosy; Active-case finding; Cluster stepped-wedge; Clinical trial; Brazil
MeSH Terms: conditions — Leprosy

STUDY DESIGN:
Intervention Model Description: Cluster stepped-wedge
Masking Description: Data analyst (statistician)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multifaceted intervention (Experimental): Implementation of active-case finding strategies
  Interventions: Other: Implementing active-case finding strategies
- Standard of care (No Intervention): Routine screening

INTERVENTIONS:
Other: Implementing active-case finding strategies — Implementation of a multifactorial active-case finding strategy, including: (1) raising awareness among the population about leprosy; (2) theoretical and practical educational training for healthcare workers; (3) georeferencing of historical and existing cases in the municipality (from 2012 to 2023) and of new cases diagnosed throughout the study (dynamic changes); (4) screening tools for signs/symptoms of the disease (application of Leprosy Suspicion Questionnaire); and (5) serological profile (rapid test) of patients with reported signs/symptoms (positive answers Leprosy Suspicion Questionnaire).
  Arms: Multifaceted intervention

SUMMARY:
The goal of this clinical trial is to assess whether a multifactorial active case-finding strategy improves the detection of leprosy cases in Brazil compared to usual screening practices. The main questions it aims to answer are:

- Does the intervention increase the number of new leprosy cases detected compared to standard care?

Participants will:

* Receive community awareness about leprosy.
* Be screened using the Leprosy Suspicion Questionnaire at priority areas identified by georeference tools.
* Undergo clinical evaluation by a trained medical team.
* If leprosy is diagnosed, affected patients will collect complementary laboratory exams

Healthcare professionals from primary care units will receive training in leprosy, while researchers will monitor changes in leprosy incidence over a 12-month period using data from Brazil's national notification system. The study will provide insights into underdiagnosis and the clinical profiles of patients who have been diagnosed.

ELIGIBILITY:
Inclusion Criteria:

(I) Municipalities

* Municipality recognized by the Brazilian Institute of Geography and Statistics as part of the Brazilian Federation.
* Municipality with operational epidemiological classification by the Ministry of Health (BMoH) as: 'municipalities with cases in the period from 2015 to 2019'.
* Municipality with authorization/consent from the government to participate in the study.

(II) Primary Health Units (Unidade Básica de Saúde or UBS) • UBS with territorial coverage (linked population) within the participating municipality.

(III) Participants

• Patients with positive Leprosy Suspicion Questionnaire (LSQ): children under five years old with Free and Informed Consent Form (ICF) signed by parents/guardians, 5-17 years old with ICF signed by parents/guardians and Free and Informed Assent Form (IAF) signed by the minor, and patients over 18 years old with ICF signed for: rapid test collection, comorbidity questionnaire and clinical evaluation; and if leprosy diagnosis is confirmed, collection of complementary exams.

Exclusion Criteria:

(I) Municipalities

* Municipality with extreme population size (municipalities with a number of inhabitants lower than the 10th percentile and higher than the 90th percentile).
* Municipality with operational epidemiological classification by the BMoH as: 'municipalities without cases in the period 2015 to 2019'.
* Municipalities with active or recent participation (less than one year) in other active-finding strategies, in addition to the usual ones: ministerial, Non-Governmental Organizations (NGOs), academic, among others.

(II) Primary Health Units

* UBS with limited multidisciplinary team (absence of physicians, nurse and/or community health agents).
* UBS with difficult access (no access by land, i.e. riverside populations).
* UBS with territorial coverage exclusively of indigenous populations.

(III) Participants

* LSQ negative.
* Patients with a previous diagnosis or history of treated leprosy.
* Patients residing/registered outside the selected municipality.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1925 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
New cases of leprosy | From the date of identification of at least one positive response in the Leprosy Suspicion Questionnaire until the date of confirmation or ruling out leprosy, assessed up to 2 months.
  Number of new cases of leprosy: incidence rate of leprosy per 100,000 inhabitants.

SECONDARY OUTCOMES:
Leprosy Suspicion Questionnaire usefulness | From the application date of the Leprosy Suspicion Questionnaire and the rapid test until the date of confirmation or ruling out leprosy, it is assessed for up to 2 months.
  Estimation of the diagnostic utility of positive LSQ and positive LSQ plus rapid test

CONTACTS AND LOCATIONS:
Overall Officials: Rosa C Lucchetta, PhD, Study Director — Hospital Alemão Oswaldo Cruz
Locations (1):
- Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR